CLINICAL TRIAL: NCT04194216
Title: Comparison of Outcomes in Rhinoplasty With the Use of Intraoperative Versus Postoperative Antibiotics
Brief Title: Antibiotic Prophylaxis in Rhinoplasty
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Washington University School of Medicine (Other); Vanderbilt University School of Medicine (Other); University of Washington (Other); Duke University (Other); Harvard University (Other); University of Kansas Medical Center (Other); University of Cincinnati (Other); Loma Linda University (Other)
Responsible Party: Principal Investigator, Sam P. Most, Professor and Chief, Division of Facial Plastic and Reconstructive Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53854
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Nasal Obstruction; Nasal Surgical Procedures
Keywords: Rhinoplasty; Antibiotic prophylaxis
MeSH Terms: conditions — Nasal Obstruction | interventions — Clindamycin; Cephalexin

STUDY DESIGN:
Intervention Model Description: Applicable Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment arm A (Active Comparator): Intra-operative single intravenous(iv) dose of "cephalexin" 2 g or "clindamycin" 900 mg.
  Interventions: Drug: Intra-operative single intravenous(iv) dose of "cephalexin" 2 g or "clindamycin" 900 mg.
- Treatment arm B (Active Comparator): Intra-operative single intravenous(iv) dose of "cephalexin" 2 g or "clindamycin" 900 mg and postoperative oral dose of "cephalexin" 250mg every 4 hours or "clindamycin" 150mg every 6 hours, for a duration of three days.
  Interventions: Drug: Intra-operative single dose (iv) of "cephalexin" 2 g or "clindamycin" 900 mg and postoperative oral dose of "cephalexin" 250mg (every 4 hours) or "clindamycin" 150mg(every 6 hours) for 3 days

INTERVENTIONS:
Drug: Intra-operative single intravenous(iv) dose of "cephalexin" 2 g or "clindamycin" 900 mg. — Treatment Arm A
  Other Names: kelfex (cephalexin); cleocin (clindamycin)
  Arms: Treatment arm A
Drug: Intra-operative single dose (iv) of "cephalexin" 2 g or "clindamycin" 900 mg and postoperative oral dose of "cephalexin" 250mg (every 4 hours) or "clindamycin" 150mg(every 6 hours) for 3 days — Treatment Arm B
  Other Names: kelfex (cephalexin); cleocin (clindamycin)
  Arms: Treatment arm B

SUMMARY:
This study compares the efficacy of a single intra-operative (intravenous) dose of "cephalexin" (first generation cephalosporin) or "clindamycin" (lincosamides), alone versus both intra-operative (intravenous) dose of "cephalexin" (first generation cephalosporin) or "clindamycin" (lincosamides) and postoperative oral dose of "cephalexin" or "clindamycin" use in nasal surgery.

DETAILED DESCRIPTION:
The study will consist of 2 treatment arms:

Treatment arm A: Intra-operative single intravenous(iv) dose of "cephalexin" 2 g or "clindamycin" 900 mg.

Treatment arm B: Intra-operative single intravenous(iv) dose of "cephalexin" 2 g or "clindamycin" 900 mg and postoperative oral dose of "cephalexin" 250mg every 4 hours or "clindamycin" 150mg every 6 hours, for a duration of three days.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (aged 18years and older)

Exclusion Criteria:

* Prior rhinoplasty
* Any exogenous (non-nasal) grafts/implants
* Immune deficiency (DM, meds, other)
* History of radiotherapy to nose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative Infection Rate | Seven days
  Postoperatively, infection rates between treatment arms will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Sam P Most, MD, Principal Investigator — Stanford Facial Plastic and Reconstructive Surgery
Locations (1):
- Facial Plastic and Reconstructive Surgery Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nuyen B, Kandathil CK, Laimi K, Rudy SF, Most SP, Saltychev M. Evaluation of Antibiotic Prophylaxis in Rhinoplasty: A Systematic Review and Meta-analysis. JAMA Facial Plast Surg. 2019 Jan 1;21(1):12-17. doi: 10.1001/jamafacial.2018.1187. PMID 30489601
- [Background] Ishii LE, Tollefson TT, Basura GJ, Rosenfeld RM, Abramson PJ, Chaiet SR, Davis KS, Doghramji K, Farrior EH, Finestone SA, Ishman SL, Murphy RX Jr, Park JG, Setzen M, Strike DJ, Walsh SA, Warner JP, Nnacheta LC. Clinical Practice Guideline: Improving Nasal Form and Function after Rhinoplasty Executive Summary. Otolaryngol Head Neck Surg. 2017 Feb;156(2):205-219. doi: 10.1177/0194599816683156. PMID 28145848
- [Background] Olds C, Spataro E, Li K, Kandathil C, Most SP. Postoperative Antibiotic Use Among Patients Undergoing Functional Facial Plastic and Reconstructive Surgery. JAMA Facial Plast Surg. 2019 Dec 1;21(6):491-497. doi: 10.1001/jamafacial.2019.1027. PMID 31647506